CLINICAL TRIAL: NCT01057186
Title: Hypophosphatemic Rickets in Norway
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 21922
Record Dates: First submitted 2010-01-26; First posted 2010-01-27 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: Hypophosphatemia, Familial; Rickets; Hyperphosphatemia
MeSH Terms: conditions — Hypophosphatemia, Familial; Rickets; Hyperphosphatemia | interventions — alfacalcidol; Phosphates; Sevelamer

STUDY DESIGN:
Observational Model: Cohort
Biospecimen Retention: Samples With DNA — EDTA plasma, serum, urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- hereditary hypophosphatemia: Norwegian patients with hereditary hypophosphatemia.
  Interventions: Dietary Supplement: Alfacalcidol; phosphate.
- Hereditary hyperphosphatemia: Norwegian patients with hereditary hyperphosphatemia (hyperphosphatemic familial tumoral calcinosis and hyperphosphatemia hyperostosis syndrome).
  Interventions: Drug: Sevelamer

INTERVENTIONS:
Dietary Supplement: Alfacalcidol; phosphate. — Individual dosage form and dosage depending on phenotype and underlying cause.
  Groups: hereditary hypophosphatemia
Drug: Sevelamer — Pills. Individual dosage depending on clinical symptoms/phenotype.
  Groups: Hereditary hyperphosphatemia

SUMMARY:
The purpose of the study is to do a follow-up survey of all individuals with hereditary hypophosphatemia in Norway, focusing on manifestations in childhood and adolescence. The investigators also want to study phenotype-genotype associations, and look for new genes, in all forms of hereditary hypo and hyperphosphatemia.

ELIGIBILITY:
Inclusion Criteria:

* All patients in the Norwegian population with hereditary hypophosphatemia, with or without rickets
* Patients in the Norwegian population with hereditary hyperphosphatemia

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The cohorts will be selected from Norwegian patients with hypophosphatemia and hyperphosphatemia.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2009-12; Primary Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Growth | Up to 18 years
  Change i height z-score from time of diagnosis to last registered consultation.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Bjerknes, Professor, MD, PhD, Study Director — Haukeland University Hospital, Pediatric department
Locations (1):
- Haukeland University Hospital, Childrens departement, Bergen, Norway